CLINICAL TRIAL: NCT06245278
Title: The Effect of Non-Surgical Periodontal Therapy on Serum And Salivary Biomarker Levels in Individuals With Inflammatory Bowel Disease
Brief Title: The Effect of Non-Surgical Periodontal Therapy on Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Profesor, Biruni University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-KAEK-80-23-03
Record Dates: First submitted 2024-01-26; First posted 2024-02-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-02

CONDITIONS: Periodontitis; Inflammatory Bowel Diseases
Keywords: Periodontitis; Inflammatory bowel disease; Cytokine
MeSH Terms: conditions — Periodontitis; Inflammatory Bowel Diseases | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clinical Healthy (Experimental): Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) salivary sample and serum will be taken from all individuals at the beginning of the study. TIM-3 levels will be examined to evaluate before and after treatment in periodontal health and periodontitis. A pre-treatment saliva sample and serum will be collected from the clinically healthy group.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)
- Periodontitis (Experimental): Non-surgical periodontal treatment will be applied to individuals with periodontitis, clinical measurements, saliva collection and serum will be repeated 12 weeks after the treatment. TIM-3 analysis will be performed by ELISA in saliva and serum of individuals. TIM-3 levels will be examined to evaluate before and after treatment in periodontal health and periodontitis. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)
- Periodontitis with İnflammatory Bowel Disease (Experimental): Non-surgical periodontal treatment will be applied to individuals with periodontitis, clinical measurements, saliva collection and serum will be repeated 12 weeks after the treatment. TIM-3 analysis will be performed by ELISA in saliva and serum of individuals. TIM-3 levels will be examined to evaluate before and after treatment in periodontitis with İnflammatory Bowel Disease. Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)
- Healthy individuals with İnflammatory Bowel Disease (Experimental): Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) salivary sample and serum will be taken from all individuals at the beginning of the study. TIM-3 levels will be examined to evaluate before and after treatment in periodontal health and periodontitis. A pre-treatment saliva sample and serum will be collected from the healthy individuals with İnflammatory Bowel Disease group.
  Interventions: Other: ELISA (Enzyme-Linked ImmunoSorbent Assay)

INTERVENTIONS:
Other: ELISA (Enzyme-Linked ImmunoSorbent Assay) — A total of 60 individuals, 15 with IBD and periodontitis, 15 with IBD and periodontal health, 15 with systemic health and periodontitis, and 15 with systemic and periodontal health, will be included in the study. At the beginning of the study, periodontal clinical measurements (gingival index, plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and serum, saliva and gingival samples will be obtained from all individuals. Individuals with periodontitis will receive non-surgical periodontal treatment in half jaws within 2 weeks. Clinical measurements, serum and saliva sample collection will be repeated 3 months after the treatment. Biomarker levels in serum and saliva samples will be analysed by ELISA.

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic and recurrent inflammatory disease of the gastrointestinal tract characterised by complex interactions between genetic susceptibility, environmental factors, microbiota and host immune response. It has two main forms, Crohn's disease (CD) and Ulcerative colitis (UC). The main mechanism of IBD pathogenesis is dysregulated host immune response to commensal microbiota and disruption of the balance of pro- and anti-inflammatory cytokines in genetically predisposed individuals. Periodontitis is a multifactorial inflammatory disease associated with dental biofilm resulting in the loss of periodontal supporting tissues and subsequently teeth. Although the occurrence of the disease depends on multifactorial factors, bacterial plaque is the primary etiological factor and various bacterial species found in plaque are responsible for initiating and maintaining the inflammatory and immune response in periodontal disease. Periodontal diseases are known to contribute to many systemic diseases/conditions or systemic disorders are known to affect periodontal disease. Although the relationship between IBD and periodontitis is based on the potential link between oral and intestinal microbiomes and host immunoinflammatory response, the pathological interactions between the two diseases have not yet been determined. From this point of view, the aim of our study was to investigate the effect of periodontal status on serum, saliva and gingival biomarkers (TIM-3, TNF-α, IL-6 and IL-17) in patients with IBD and to evaluate the relationship between these values and periodontal clinical parameters. This is the first study to examine TIM-3 levels in saliva, serum and gingival samples in patients with IBD and periodontitis with IBD.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65,
* Having at least 8 teeth excluding wisdom teeth,
* No periodontal treatment in the last 3 months,
* Not having used antibiotics in the last 3 months,
* Not being pregnant or breastfeeding,
* The individuals to be included in the control group should not have any systemic disease that may change the periodontal status, and the individuals to be included in the experimental group should not have any systemic disease that may affect periodontal health except IBD.

Exclusion Criteria:

* Under 18 years of age and over 65 years of age,
* Having less than 8 teeth,
* Having undergone periodontal treatment in the last 3 months,
* Having used antibiotics in the last 3 months,
* Being pregnant or breastfeeding,
* Individuals to be included in the control group should have any systemic disease that may change the periodontal status, and individuals to be included in the test group should have any systemic disease that may affect periodontal health except IBD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Examination of TIM-3 levels of periodontal disease and inflammatory bowel disease | up to 1 year
  Examination of TIM-3 levels, which are stated to be associated with periodontal disease, in serum and saliva samples obtained from individuals with periodontitis and periodontitis individuals with inflammatory bowel disease.

SECONDARY OUTCOMES:
Evaluation of the effect of non-surgical periodontal treatment on changes in TIM-3 level. | up to 1 year
  Evaluation of the effect of non-surgical periodontal treatment on changes in TIM-3 level.

OTHER OUTCOMES:
Comparison biomarkers of study groups. | up to 1 year
  Comparison of serum and saliva samples taken before treatment in individuals with periodontitis and periodontitis individuals with inflammatory bowel disease in terms of TIM-3 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No